CLINICAL TRIAL: NCT01349036
Title: A Phase 2 Study of Orally Administered PLX3397 in Patients With Recurrent Glioblastoma
Brief Title: A Phase 2 Study of PLX3397 in Patients With Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-04
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Glioblastoma
Keywords: Glioblastoma; brain cancer
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLX3397-Cohort 1 (Experimental): 10 patients with recurrent glioblastoma who require reoperation will be treated with PLX3397 for 7 days prior to surgery and their tumor tissue will be evaluated for pharmacokinetic levels and pharmacodynamic effects.
  Interventions: Drug: PLX3397
- PLX3397-Cohort 2 (Experimental): 30 patients will be orally dosed with PLX3397 continuously on 28 day cycles.
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Capsules administered once or twice daily, continuous dosing
  Other Names: Pexidartinib

SUMMARY:
The objective of this study is to evaluate the response of subjects with recurrent glioblastoma to continuous therapy of PLX3397.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old with a life expectancy of at least 8 weeks
* Radiographically proven recurrent (≥ first relapse), intracranial Glioblastoma (GBM)
* For all patients, availability of at least 10 unstained slides (or archival tumor block sufficient to generate at least 10 unstained slides) from any previous GBM surgery
* Previous treatment with external beam radiation and temozolomide chemotherapy
* Before the first dose of PLX3397,adequate recovery from toxicity of prior therapy as follows:

>28 days for cytotoxic therapy >42 days for nitrosoureas >28 days for bevacizumab >7 days for non cytotoxic therapy such as interferon, tamoxifen, thalidomide, cis-retinoic acid, or erlotinib

* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use an acceptable method of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year. Men of child-bearing potential must also agree to use an acceptable method of birth control while on study drug.
* Karnofsky performance status of ≥60
* Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥1.0 x 109/L, Hgb >9 g/dL, platelet count ≥50 x 109/L, Aspartate aminotransferase/Alanine aminotransferase (AST/ALT) ≤2.5x Upper Limit of Normal (ULN), creatinine ≤1.5x ULN)
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements

Exclusion Criteria:

* Investigational drug use within 28 days of the first dose of PLX3397
* GBM progression within 3 months of previous radiation by Response Assessment in Neuro-Oncology (RANO) criteria
* History of Grade 2 Common Toxicity Criteria for Adverse Events (CTCAE v4) or greater acute intracranial hemorrhage
* Previous failure of bevacizumab or other vascular endothelial growth factor (VEGF) therapy except in a first line setting
* History of malignant glioma with co-deletion of 1p/19q
* A concurrent active cancer that requires non-surgical therapy (e.g. chemotherapy, radiation, adjuvant therapy). Prior history of other cancer is allowed, as long as there was no active disease within the prior 3 years.
* Refractory nausea and vomiting, malabsorption, biliary shunt, or significant bowel resection that would preclude adequate absorption
* Patients with serious illnesses, uncontrolled infection, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
* Women of child-bearing potential who are pregnant or breast feeding
* corrected QT interval (QTc) ≥450 msec at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-12-03 (Actual); Primary Completion 2013-11-05 (Actual); Study Completion 2013-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University California, Los Angeles, Los Angeles, California
  - University California, San Francisco, San Francisco, California
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Lamborn KR, Yung WK, Chang SM, Wen PY, Cloughesy TF, DeAngelis LM, Robins HI, Lieberman FS, Fine HA, Fink KL, Junck L, Abrey L, Gilbert MR, Mehta M, Kuhn JG, Aldape KD, Hibberts J, Peterson PM, Prados MD; North American Brain Tumor Consortium. Progression-free survival: an important end point in evaluating therapy for recurrent high-grade gliomas. Neuro Oncol. 2008 Apr;10(2):162-70. doi: 10.1215/15228517-2007-062. Epub 2008 Mar 4. PMID 18356283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 38 participants who met all inclusion and none of the exclusion criteria were enrolled and received the study drug.
Pre-assignment Details: Enrollment planned to include approximately 40 participants (10 in Cohort 1 and 30 in Cohort 2) recruited from approximately 6 clinic sites.
Groups:
- PLX3397 - Cohort 1 (Surgical): Participants with recurrent glioblastoma who required reoperation were treated with PLX3397 for 7 days prior to surgery.
- PLX3397 - Cohort 2 (Non-surgical): Participants who received PLX3397 continuously on 28 day cycles.
Period: Overall Study
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Started | 14 | 24
Completed | 0 | 0
Not Completed | 14 | 24
Not completed — Disease progression | 13 | 22
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PLX3397 - Cohort 2 (Non-surgical): Participants with recurrent glioblastoma who received PLX3397 continuously on 28 day cycles.
- Total: Total of all reporting groups
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical) | Total
Number analyzed (Participants) | 14 | 24 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (8.6) | 54.1 (11.7) | 54.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 17 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 21 | 35
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 24 | 38

OUTCOME MEASURES:

1. Primary Outcome: Summary of Response Rates in Participants on Treatment With PLX3397
Description: Response to treatment was evaluated using the Response Assessment in Neuro-Oncology (RANO) criteria. All participants were evaluated for progression free survival (PFS), and overall survival (OS). The six-month PFS rate was defined as the number of subjects with PFS of at least 6-month duration, with PFS measured from the first day of treatment (Cycle 1, Day 1) to the date of the first documented disease progression or date of death, whichever occurs first, over a 6-month period and evaluated using the Kaplan Meier method. The rate of OS was defined as the number of subjects that survived until study exit.
Time Frame: 6 months post dose
Population: Response rates were assessed in the modified intent-to-treat population.
Measure: Count of Participants; unit: Participants
Groups:
- Surgical Cohort 1 (N=14): Participants with recurrent glioblastoma who were treated with PLX3397 in Cohort 1 (surgical).
- Non-Surgical Cohort 2 (N=24): Participants with recurrent glioblastoma who were treated with PLX3397 in Cohort 2 (non-surgical).
Arm/Group | Surgical Cohort 1 (N=14) | Non-Surgical Cohort 2 (N=24)
Number analyzed (Participants) | 13 | 22
Participants
  Six-month PFS rate | 1 | 2
  Overall survival | 10 | 21
  Complete response rate | 0 | 0
  Partial response rate | 0 | 0
  Stable disease rate | 3 | 4
  Progressive disease rate | 10 | 18
  Not Evaluable | 1 | 2

2. Primary Outcome: Mean Plasma Pharmacokinetic Parameters of PLX3397 After Oral Administration of 1000 mg/Day - Cycle 1 Day 15
Description: A noncompartmental method of analysis was used to analyze the plasma concentrations of PLX3397. Mean plasma pharmacokinetic parameters, include time to maximum concentration (Tmax) and will be calculated from the Cycle 1, Day 15 values.
Time Frame: Pre-dose and up to 6 post dose during cycle 1, Day 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Number analyzed (Participants) | 11 | 21
hours | 2.09 (1.04) | 1.71 (0.90)

3. Primary Outcome: Mean Plasma Pharmacokinetic Parameters of PLX3397 After Oral Administration of 1000 mg/Day - Cycle 1 Day 15
Description: A noncompartmental method of analysis was used to analyze the plasma concentrations of PLX3397. Mean plasma pharmacokinetic parameters include maximum concentration (Cmax) and will be calculated from the Cycle 1, Day 15 values.
Time Frame: Pre-dose and up to 6 post dose during cycle 1, Day 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Number analyzed (Participants) | 11 | 21
ng/mL | 7760 (2330) | 8030 (2790)

4. Primary Outcome: Mean Plasma Pharmacokinetic Parameters of PLX3397 After Oral Administration of 1000 mg/Day - Cycle 1 Day 15
Description: A noncompartmental method of analysis was used to analyze the plasma concentrations of PLX3397. Mean plasma pharmacokinetic parameters include an assessment of area under the curve over 0-4 hours (AUC0-4), and will be calculated from the Cycle 1, Day 15 values.
Time Frame: Pre-dose and up to 6 post dose during cycle 1, Day 15
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Number analyzed (Participants) | 11 | 21
hr*ng/mL | 24900 (6700) | 26100 (9260)

5. Primary Outcome: Mean Plasma Pharmacokinetic Parameters of PLX3397 After Oral Administration of 1000 mg/Day - Cycle 1 Day 15
Description: A noncompartmental method of analysis was used to analyze the plasma concentrations of PLX3397. Mean plasma pharmacokinetic parameters include an assessment of area under the curve over 0-6 hours (AUC0-6), and will be calculated from the Cycle 1, Day 15 values.
Time Frame: Pre-dose and up to 6 post dose during cycle 1, Day 15
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Number analyzed (Participants) | 11 | 21
hr*ng/mL | 36100 (10000) | 36900 (12200)

6. Secondary Outcome: Incidence (Number and Percentage of Participants) With Treatment-Emergent Adverse Events Related to Study Drug Occurring in ≥10% Participants During Treatment With PLX3397 (Safety Population)
Time Frame: Up to 1 year post dose
Population: Safety events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- PLX3397 - Cohort 1 (Surgical): All participants with recurrent glioblastoma who were treated with PLX3397 in Cohort 1 (surgical).
- PLX3397 - Cohort 2 (Non-surgical): All participants with recurrent glioblastoma who were treated with PLX3397 in Cohort 2 (non-surgical).
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
Number analyzed (Participants) | 14 | 24
Participants
  Any Event | 12 | 22
  Fatigue | 6 | 14
  Constipation | 3 | 1
  Nausea | 1 | 3
  Hair color changes | 2 | 4
  Aspartate aminotransferase increased | 3 | 3
  Alanine aminotransferase increased | 2 | 3
  Decreased appetite | 3 | 3
  Headache | 1 | 3
  Pyrexia | 2 | 1
  Dry Mouth | 2 | 0
  Rash | 2 | 1
  Neutropenia | 0 | 3
  Lymphopenia | 2 | 0
  Blood Lactate Dehydrogenase Increased | 2 | 1
  Hypertension | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from after the first dose to 28 days after the last dose.
Description: Adverse events that emerge (or worsen) after the first dose of study drug and within 28 days after the last dose.
Arm/Group | PLX3397 - Cohort 1 (Surgical) | PLX3397 - Cohort 2 (Non-surgical)
All-Cause Mortality (participants affected / at risk) | 0/14 | 1/24
Serious Adverse Events (participants affected / at risk) | 8/14 | 11/24
Other Adverse Events (participants affected / at risk) | 14/14 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 - Cohort 1 (Surgical) (N=14) | PLX3397 - Cohort 2 (Non-surgical) (N=24)
Convulsion (Nervous system disorders) | 3 | 5
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
ALT increased (Investigations) | 0 | 1
AST increased (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 1
WBC count decreased (Investigations) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 - Cohort 1 (Surgical) (N=14) | PLX3397 - Cohort 2 (Non-surgical) (N=24)
Headache (Nervous system disorders) | 6 | 8
Convulsion (Nervous system disorders) | 4 | 4
Dizziness (Nervous system disorders) | 5 | 2
Hemiparesis (Nervous system disorders) | 2 | 3
Aphasia (Nervous system disorders) | 3 | 1
Memory impairment (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 1 | 2
Hemianopia (Nervous system disorders) | 2 | 1
Psychomotor skills impaired (Nervous system disorders) | 1 | 2
Ataxia (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 2 | 0
Dyaesthesia (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 7 | 14
Pyrexia (General disorders) | 5 | 2
Gait disturbance (General disorders) | 2 | 2
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 2
Lacrimation increased (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 1 | 1
Diplopia (Eye disorders) | 1 | 0
Eye disorder (Eye disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 6
Deep vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Candidiasis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Skin candida (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 3
Alanine aminotransferase increased (Investigations) | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 2
Blood albumin decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Incision site pain (Injury, poisoning and procedural complications) | 2 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 3
Micturition urgency (Injury, poisoning and procedural complications) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was terminated due to results noted in primary outcome measure 1. The sponsor felt that the PFS 6 goal of 25% (Lamborn, 2008) was unlikely to be met upon further enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No